CLINICAL TRIAL: NCT02283164
Title: Randomized Controlled Trial to Improve Oncology Nurses' Protective Equipment Use
Brief Title: Drug Exposure Feedback and Education for Nurses' Safety
Acronym: DEFENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher R. Friese, Elizabeth Tone Hosmer Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HUM00103873
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Occupational Health; Hazardous Material Handling
Keywords: Occupational health; Hazardous material handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Hazardous materials online education and study feedback
  Interventions: Behavioral: Hazardous materials online education and study feedback
- Control then treatment (Active Comparator): Hazardous materials online education and study feedback
  Interventions: Behavioral: Hazardous materials online education and study feedback

INTERVENTIONS:
Behavioral: Hazardous materials online education and study feedback — Participants will receive a 45-minute educational webinar on hazardous materials handing best practices at the beginning of the intervention period. Subsequently they will receive quarterly feedback of interim study results.

SUMMARY:
The goal of this research is to evaluate the efficacy of an audit and feedback intervention to improve personal protective equipment (PPE) use by nurses who handle hazardous drugs in the ambulatory oncology setting.

DETAILED DESCRIPTION:
The overall objective of the proposed study is to investigate exposures to hazardous antineoplastic drugs among oncology nurses who handle them. The specific project objective is to evaluate the efficacy of an audit and feedback intervention to improve PPE use by nurses who handle hazardous drugs in the ambulatory oncology setting. This project will pursue three specific aims:

1. Evaluate the efficacy of an audit and feedback intervention to improve recommended use of PPE;
2. Determine whether the intervention effects on PPE use are mediated by knowledge about PPE use and perceived risk of hazardous drug exposure, and;
3. Determine whether the intervention effects on PPE use are moderated by personal (experience, education, certification) and organizational factors (workloads, practice environments, safety organizing).

To achieve these aims, 382 nurses employed in 11 oncology centers will participate in a cluster randomized controlled trial. Sites will be randomized so participants will receive a one-hour web-based educational module on hazardous drug safe handling with quarterly email reminders about the educational content (control) or the web-based educational module plus quarterly feedback on hazardous drug spills and drug levels measured in the study population (treatment). The hypothesis is that nurses in sites who receive the treatment will report significantly higher PPE use compared to nurses in sites assigned to receive the control. Data will also identify organizational factors that can be targeted for future interventions.

ELIGIBILITY:
Inclusion Criteria:

* registered nurses
* employed 16 hours or more per week in the ambulatory chemotherapy infusion area

Exclusion Criteria:

* Treatment with an antineoplastic agent in the past year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Usage of PPE | Baseline (Year 1) and follow-up (Year 3)
  Use of PPE is measured on a 6-point Likert scale (5=always, 4=76-99% of the time, 3=51-75%, 2=26-50%, 1=1-25%, and 0=never). A mean score is calculated for each participant across 5 items: use of chemotherapy gloves, double gloves, single-use disposable gowns, eye protection, and respirators. Higher scores reflect more frequent use of PPE elements.

SECONDARY OUTCOMES:
Potential Mediators | Baseline (Year 1) and follow-up (Year 3)
  Knowledge of PPE and perceived risk of hazardous drug exposure are hypothesized to mediate the potential effects of the intervention on PPE use.
  1. Knowledge of PPE will be measured using a 10-item chemotherapy exposure knowledge scale. Individual questions about drug exposure are multiple choice. Correct answers are scored as 1 and incorrect answers are scored as 0. The scale range is 0-10, with higher scores reflecting increased knowledge.
  2. Perceived risk of drug exposure will be measured using a 3-item subscale from Geer's Occupational Dermal Survey. A 4-point Likert scale (1=strongly disagree, 4=strongly agree) will be used to assess nurses' perceptions of the risks of chemotherapy exposure and potential health effects
Potential Moderators--Organization | Baseline (Year 1) and follow-up (Year 3)
  Three organizational factors (workloads, practice environments, and safety organizing) are proposed moderators:
  1. Workloads will be measured by the number of patients participants had primary responsibility for on their last shift.
  2. The practice environment will be measured by calculating the average of a 23-item composite measure across six domains: nurse participation in practice affairs, nursing foundations for quality care, nurse manager support and leadership, collegial nurse-physician relations, staffing and resource adequacy, and medical assistant support. Items are scored on a 5-point Likert scale, where 1=strongly disagree to 5=strongly agree the characteristic is present in the practice.
  3. The Safety Organizing Scale (SOS) reflects theoretically derived and empirically observed content domains in high-reliability organizations that avert operational failure. Each item is scored on a 7-point Likert scale (1=not at all, 7=to a very great extent).
Potential Moderators--Personal | Baseline (Year 1) and follow-up (Year 3)
  Three personal factors (experience, education, and certification) are proposed moderators.
  1. nursing experience (years),
  2. education (diploma, associate's degree, bachelor's degree, master's degree, post-master's degree)
  3. certification (Oncology Nursing Society chemotherapy certification, Oncology Certified Nurse (OCN®), Advanced Oncology Certified Nurse (AOCN®), other certification)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Friese, PhD, Principal Investigator — University of Michigan School of Nursing

REFERENCES:
- [Background] Friese CR, Mendelsohn-Victor K, Wen B, Sun D, Sutcliffe K, Yang JJ, Ronis DL, McCullagh MC; DEFENS Study Investigators. DEFENS - Drug Exposure Feedback and Education for Nurses' Safety: study protocol for a randomized controlled trial. Trials. 2015 Apr 17;16:171. doi: 10.1186/s13063-015-0674-5. PMID 25928792
- [Background] Friese CR, Yang J, Mendelsohn-Victor K, McCullagh M. Randomized Controlled Trial of an Intervention to Improve Nurses' Hazardous Drug Handling. Oncol Nurs Forum. 2019 Mar 1;46(2):248-256. doi: 10.1188/19.ONF.248-256. PMID 30767961